CLINICAL TRIAL: NCT04550065
Title: SMART Family-Link Project: A Digital Game on Promoting Family Well-being
Brief Title: A Digital Game on Promoting Family Well-being
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW 20-353
Record Dates: First submitted 2020-09-07; First posted 2020-09-16 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Family
Keywords: Family well-being; Family communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Digital game
  Interventions: Behavioral: Digital game

INTERVENTIONS:
Behavioral: Digital game — A digital family game with theme-based mini games (epidemic prevention, exercise, diet, communication and parenting)

SUMMARY:
Advances in information communication technologies (ICT) allow for ICT-assisted health promotion to become more common. Integrating ICT in health promotion has been suggested to offer many advantages compared to traditional approaches to promote family well-being. Research has also shown the positive effects of game-based approaches in enhancing health promotion interventions, especially with children. We will develop and assess a digital family game with theme-based mini-games to enhance family communication and well-being.

DETAILED DESCRIPTION:
With growing emphasis on the development and maintenance of healthy lifestyles, the family role has increasing importance. A family-based health promotion strategy can be instrumental in helping disseminate and reinforce knowledge and behaviours on family well-being and better equip families to protect themselves and promote family well-being amidst the pandemic.

This study aims to use a game-based approach to enhance knowledge and behaviours on family well-being. We will conduct quantitative and qualitative evaluation. The findings would provide preliminary evidence of the feasibility and effectiveness of such an approach in a family-based context. It would also guide the direction for future health education and awareness trials and related projects and campaigns for health promotion efforts and to help improve family well-being in the Hong Kong community and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Chinese-speaking;
* Individuals aged 18 years and above;
* Able to understand and play the game.

Exclusion Criteria:

* Individuals who cannot meet the inclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Perceived improved family well-being | Baseline and one month
  Change assessed by a validated one-item Family Happiness scale (score from 0 to 10, higher scores indicate more family happiness).

SECONDARY OUTCOMES:
Perceived improved family communication | Baseline and one month
  Change assessed by a one-item family communication scale (score from 0 to 10, higher scores indicate better family communication).
Perceived improved family health | Baseline and one month
  Change assessed by a one-item family health scale (score from 0 to 10, higher scores indicate better family health).
Family well-being knowledge and behaviors | Baseline and one month
  Change assessed by outcome-based questions (scores from 0 to 10, higher scores indicate better knowledge and behaviors)
Practice of sharing family well-being knowledge | One month
  Assessed by outcome-based questions with categorical choices

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Y Lai, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Hong Kong community, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Will share after study finished
Supporting Information: Study Protocol
Time Frame: Baseline and 1 month
Access Criteria: The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact, Ms Shirley Sit (email shirlsit@hku.hk), (School of Public Health, The University of Hong Kong) for further information.

REFERENCES:
- [Background] Ameryoun A, Sanaeinasab H, Saffari M, Koenig HG. Impact of Game-Based Health Promotion Programs on Body Mass Index in Overweight/Obese Children and Adolescents: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Child Obes. 2018 Feb/Mar;14(2):67-80. doi: 10.1089/chi.2017.0250. Epub 2017 Nov 29. PMID 29185787
- [Background] Chagas CMDS, Pontes E Silva TB, Reffatti LM, Botelho RBA, Toral N. Rango Cards, a digital game designed to promote a healthy diet: a randomized study protocol. BMC Public Health. 2018 Jul 24;18(1):910. doi: 10.1186/s12889-018-5848-0. PMID 30041639
- [Background] Edwards EA, Lumsden J, Rivas C, Steed L, Edwards LA, Thiyagarajan A, Sohanpal R, Caton H, Griffiths CJ, Munafo MR, Taylor S, Walton RT. Gamification for health promotion: systematic review of behaviour change techniques in smartphone apps. BMJ Open. 2016 Oct 4;6(10):e012447. doi: 10.1136/bmjopen-2016-012447. PMID 27707829
- [Derived] Sit SM, Lai AY, Wong HW, Hung KS, Wang MP, Ho SY, Lam TH. Gamified Strength Recognition and Quiz to Enhance COVID-19 Prevention, Knowledge, Behaviors, and Family Well-Being. Games Health J. 2024 Jun;13(3):172-183. doi: 10.1089/g4h.2023.0190. Epub 2024 Mar 20. PMID 38512294